CLINICAL TRIAL: NCT07302230
Title: The EMPOWER Trial: Evaluating a Home-Based Physical Activity Program (PAP) With the ExerciseRx™ Digital Platform vs. Health Education Group (HEG) in People With Non-Muscle Invasive Bladder Cancer
Brief Title: Home-Based Physical Activity Program With Digital App Versus Health Education Group for Improving Physical Activity Among Patients With Non-muscle Invasive Bladder Cancer, The EMPOWER Trial
Acronym: EMPOWER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Andy Hill CARE Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RG1125987; NCI-2025-08850 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21052 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Localized Non-Muscle Invasive Bladder Urothelial Carcinoma; Stage 0a Bladder Cancer AJCC v8; Stage 0is Bladder Cancer AJCC v8; Stage I Bladder Cancer AJCC v8
Keywords: Urinary Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Interviews as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study statistician will be blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: Health Education Group (HEG) (Active Comparator): Patients receive recommendations from their physicians to continue their usual physical activity as tolerated, receive a FitBit® to wear continuously throughout the study, with the ExerciseRx app locked to the baseline home screen, and receive an educational pamphlet describing physical activity goals in line with NCCN Survivorship for Healthy Living Guidelines.
  Interventions: Other: Best Practice; Other: Internet-Based Intervention; Other: Health Telemonitoring; Other: Educational Intervention; Other: Questionnaire Administration; Other: Interview; Other: Electronic Health Record Review
- Group II: Physical Activity Program (PAP) intervention (Experimental): Patients complete home exercise sessions given via the ExerciseRx app over 20-30 minutes 4 times per week for 12 weeks and receive daily step count goals. Patients also receive a FitBit® to wear continuously throughout the study, and are given access to view their step counts via the ExerciseRx app, and receive an educational pamphlet as in Group I.
  Interventions: Other: Internet-Based Intervention; Other: Exercise Intervention; Other: Health Telemonitoring; Other: Educational Intervention; Other: Questionnaire Administration; Other: Interview; Other: Electronic Health Record Review

INTERVENTIONS:
Other: Internet-Based Intervention — Given access to the ExerciseRx app
  Arms: Group II: Physical Activity Program (PAP) intervention
Other: Best Practice — Given instruction to continue physical activity as usual
  Other Names: standard of care
  Arms: Group I: Health Education Group (HEG)
Other: Internet-Based Intervention — Given access to the ExerciseRx app locked to the baseline home screen
  Arms: Group I: Health Education Group (HEG)
Other: Exercise Intervention — Complete home exercise sessions
  Arms: Group II: Physical Activity Program (PAP) intervention
Other: Health Telemonitoring — Given a FitBit® to wear continuously
Other: Educational Intervention — Given NCCN Survivorship for Healthy Living Guidelines pamphlet
Other: Questionnaire Administration — Ancillary studies
Other: Interview — Ancillary studies
Other: Electronic Health Record Review — Ancillary studies

SUMMARY:
This clinical trial compares how well a home-based personalized physical activity program (PAP) that is delivered by a digital application (app) (the ExerciseRx app) works compared to health education in improving physical activity for patients with bladder cancer that has not reached the muscle wall of the bladder (non-muscle invasive). For people who are not physically active, previous studies have shown that increasing step counts can reduce incidence of death, reduce frailty, and reduce healthcare costs. The ExerciseRx app tracks adherence to home exercise, adapts step count goals based on the patient's progress, and provides encouraging feedback and motivation from the healthcare team. Additional features include activity summaries, progress towards current goal, nudges, helpful facts about the benefits of activity, and ideas for how to incorporate daily movement. A home-based PAP using the ExerciseRx app may work better in increasing physical activity among patients with non-muscle invasive bladder cancer compared to a health education only group.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (Health Education Group, HEG): Patients receive recommendations from their physicians and an educational pamphlet describing physical activity goals in line with National Comprehensive Cancer Network (NCCN) Survivorship for Healthy Living Guidelines. They receive a FitBit® to wear continuously throughout the study, with the ExerciseRx app locked to the baseline home screen.

GROUP II (PAP INTERVENTION): Patients complete home exercise sessions given via the ExerciseRx app over 20-30 minutes 4 times per week for 12 weeks and receive personalized daily step count goals that gradually increase over the study period. Patients also receive a FitBit® to wear continuously throughout the study, are given access to features of the ExerciseRx app (step count goals, home exercise videos), and receive an educational pamphlet as in Group I.

After completion of the study intervention, patients are followed up at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age >= 18 years)
* Prior diagnosis of non-muscle invasive bladder cancer (NMIBC), currently on surveillance or receiving maintenance intravesical therapy (including intravesical chemotherapy, immunotherapy)
* Classified as insufficiently active on the Physical Activity as a Vital Sign (PAVS) assessment
* Has an Android or Apple Smartphone/Tablet
* Ambulatory
* English-speaking
* Willing and able to participate in study activities and sign the informed consent form

Exclusion Criteria:

* Severe cognitive or memory impairment/dementia precluding ability to follow instructions or participate in survey assessments
* Inability to read or understand English
* Lack of access or lack of sufficient facility to use an Android or iOS smart device with the minimum criteria to run the ExerciseRx app
* Not receiving treatment at University of Washington (UW)
* Orthopedic, neurologic, or other problems that prevent safe ambulation and protocol adherence. Information on prior falls and other recent orthopedic or neurologic problems will be used to make judgment about protocol eligibility
* Inability/Unwillingness to participate in a personalized exercise program
* Current diagnosis with muscle-invasive or metastatic bladder cancer
* Uncontrolled or concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Lack of access or lack of sufficient facility to use an Android or iOS smart device with the minimum criteria for using the ExerciseRx app
* Participation in a clinical trial that does not permit enrollment in the EMPOWER trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-11 (Estimated); Primary Completion 2027-02-26 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in mean daily step count | Baseline (1 week prior to trial initiation) and timepoint 2 (12 weeks)
  Average daily step count (per 24-hour day) will be assessed by the Fitbit tracker. Summary statistics (mean and standard deviations; counts and percentages) will be used to describe and compare baseline characteristics between the two treatment arms. Will use a linear mixed effects model with average daily step count as the outcome, with fixed effects for time (T1, T2, and T3), treatment assignment, and the week-treatment interaction, and a random intercept for each participant. A significant interaction between T2 and treatment assignment will indicate the change in step count from baseline to T2 differs between the two treatment arms and will be used to evaluate the co-primary outcomes of step-count improvement at the end of treatment using a two-sided significance level of 0.05. The minimum amount of time that participants need to have worn the Fitbit for their step data to be valid for use in analysis is one week (7 days) post baseline period.
Qualitative experience | Week 16
  Will be assessed by Zoom interviews (usability interview) with a subset of volunteer participants from the physical activity program (PAP) arm. Will analyze the semi-structured interview data using a process of reflexive thematic analysis, drawing on our reflexivity as designers, health informatics researchers, and clinical researchers to interpret data and construct themes using affinity analysis to identify ways in which ExerciseRx can be improved to meet the needs of patients with bladder cancer. Similarly, will apply the Discover Design Built Test framework from the University of Washington ALACRITY Center to adapt the ExerciseRx provider dashboard for healthcare providers caring for patients with bladder cancer.

SECONDARY OUTCOMES:
Active time/24 hours (minutes) per week on study | Up to 12 weeks
  A linear mixed effect model will be used to analyze the impact of the ExerciseRx platform comparing PAP to Health Education Group (HEG). Each model will include this outcome with fixed effects for time, treatment assignment, and the time-treatment interaction as well as a random effect for each participant to account for repeated measures. Significant interaction terms will indicate a treatment effect is present at that measurement time.
Change in mean daily step count | Baseline up to 4 weeks post intervention
  A linear mixed effect model will be used to analyze the impact of the ExerciseRx platform comparing PAP to HEG. Each model will include this outcome with fixed effects for time, treatment assignment, and the time-treatment interaction as well as a random effect for each participant to account for repeated measures. Significant interaction terms will indicate a treatment effect is present at that measurement time.
Change in functional mobility | Baseline up to 4 weeks post intervention
  Assessed by the Short Physical Performance Battery. A linear mixed effect model will be used to analyze the impact of the ExerciseRx platform comparing PAP to HEG. Each model will include this outcome with fixed effects for time, treatment assignment, and the time-treatment interaction as well as a random effect for each participant to account for repeated measures. Significant interaction terms will indicate a treatment effect is present at that measurement time.
Change in frailty | Baseline up to 4 weeks post intervention
  Assessed by the Cancer and Aging Research Group - Geriatric Assessment. A linear mixed effect model will be used to analyze the impact of the ExerciseRx platform comparing PAP to HEG. Each model will include this outcome with fixed effects for time, treatment assignment, and the time-treatment interaction as well as a random effect for each participant to account for repeated measures. Significant interaction terms will indicate a treatment effect is present at that measurement time.
Change in health-related quality of life | Baseline up to 4 weeks post intervention
  Will include physical function, role function, emotional function, cognitive function, and social function. Assessed by the European Organization for Research and Treatment of Cancer - Quality of Life Questionnaire (Core 30) (EORTC-QLQ-C30) and EORTC Quality of Life Questionnaire - Non-Muscle-Invasive Bladder Cancer Module (24 items) (EORTC-QLQ-NMIBC24). A linear mixed effect model will be used to analyze the impact of the ExerciseRx platform comparing PAP to HEG. Each model will include this outcome with fixed effects for time, treatment assignment, and the time-treatment interaction as well as a random effect for each participant to account for repeated measures. Significant interaction terms will indicate a treatment effect is present at that measurement time.
Change in fatigue | Baseline up to 4 weeks post intervention
  Will be assessed using the Insomnia and Symptom Scale of the EORTC-QLQ-C30. A linear mixed effect model will be used to analyze the impact of the ExerciseRx platform comparing PAP to HEG. Each model will include this outcome with fixed effects for time, treatment assignment, and the time-treatment interaction as well as a random effect for each participant to account for repeated measures. Significant interaction terms will indicate a treatment effect is present at that measurement time.
Change in pain | Baseline up to 4 weeks post intervention
  Will be assessed using the Symptom Scale of the EORTC-QLQ-C30. A linear mixed effect model will be used to analyze the impact of the ExerciseRx platform comparing PAP to HEG. Each model will include this outcome with fixed effects for time, treatment assignment, and the time-treatment interaction as well as a random effect for each participant to account for repeated measures. Significant interaction terms will indicate a treatment effect is present at that measurement time.
Change in anxiety/depression | Baseline up to 4 weeks post intervention
  Will be assessed using the Hospital Anxiety and Depression Scale (HADS)-Anxiety and HADS-Depression (14 items). A linear mixed effect model will be used to analyze the impact of the ExerciseRx platform comparing PAP to HEG. Each model will include this outcome with fixed effects for time, treatment assignment, and the time-treatment interaction as well as a random effect for each participant to account for repeated measures. Significant interaction terms will indicate a treatment effect is present at that measurement time.
Change in distress | Baseline up to 4 weeks post intervention
  Will be assessed using the Perceived Stress Scale. A linear mixed effect model will be used to analyze the impact of the ExerciseRx platform comparing PAP to HEG. Each model will include this outcome with fixed effects for time, treatment assignment, and the time-treatment interaction as well as a random effect for each participant to account for repeated measures. Significant interaction terms will indicate a treatment effect is present at that measurement time.
Change in resiliency | Baseline up to 4 weeks post intervention
  Will be assessed using the Brief Resiliency Scale. A linear mixed effect model will be used to analyze the impact of the ExerciseRx platform comparing PAP to HEG. Each model will include this outcome with fixed effects for time, treatment assignment, and the time-treatment interaction as well as a random effect for each participant to account for repeated measures. Significant interaction terms will indicate a treatment effect is present at that measurement time.
Change in treatment burden | Baseline up to 4 weeks post intervention
  Will be assessed using the Treatment Burden Questionnaire (engagement in healthcare). Each model will include this outcome with fixed effects for time, treatment assignment, and the time-treatment interaction as well as a random effect for each participant to account for repeated measures. Significant interaction terms will indicate a treatment effect is present at that measurement time.
Incidence of patient-reported musculoskeletal adverse events | Baseline up to 4 weeks post intervention
  A linear mixed effect model will be used to analyze the impact of the ExerciseRx platform comparing PAP to HEG. Each model will include this outcome with fixed effects for time, treatment assignment, and the time-treatment interaction as well as a random effect for each participant to account for repeated measures. Significant interaction terms will indicate a treatment effect is present at that measurement time.
Incidence of treatment-associated toxicity | Baseline up to 4 weeks post intervention
  Will be assessed using the EORTC-NMIBC 24. A linear mixed effect model will be used to analyze the impact of the ExerciseRx platform comparing PAP to HEG. Each model will include this outcome with fixed effects for time, treatment assignment, and the time-treatment interaction as well as a random effect for each participant to account for repeated measures. Significant interaction terms will indicate a treatment effect is present at that measurement time.
Incidence of patient-reported outcomes | Up to 4 weeks post intervention
  Will be assessed using the Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events version 5.0 and chart review. A linear mixed effect model will be used to analyze the impact of the ExerciseRx platform comparing PAP to HEG. Each model will include this outcome with fixed effects for time, treatment assignment, and the time-treatment interaction as well as a random effect for each participant to account for repeated measures. Significant interaction terms will indicate a treatment effect is present at that measurement time.
Barriers and facilitators to exercise | Baseline up to 4 weeks post intervention
  Will be assessed using the weekly barriers and facilitators to exercise survey. A linear mixed effect model will be used to analyze the impact of the ExerciseRx platform comparing PAP to HEG. Each model will include this outcome with fixed effects for time, treatment assignment, and the time-treatment interaction as well as a random effect for each participant to account for repeated measures. Significant interaction terms will indicate a treatment effect is present at that measurement time.
Change in Lifespace | Baseline up to 4 weeks post intervention
  Will be assessed using the Lifespace questionnaire. A linear mixed effect model will be used to analyze the impact of the ExerciseRx platform comparing PAP to HEG. Each model will include this outcome with fixed effects for time, treatment assignment, and the time-treatment interaction as well as a random effect for each participant to account for repeated measures. Significant interaction terms will indicate a treatment effect is present at that measurement time.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Psutka, MD, MSc, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No